CLINICAL TRIAL: NCT02087930
Title: Microbiota as Potential Target for Innovative Preventive and Therapeutic Strategies for Food Allergy
Brief Title: Microbiota as Potential Target for Food Allergy
Acronym: MATFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 02/14
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

GROUPS / COHORTS (2):
- Cow milk allergy children: Children affected by Immunoglobulin E medited cow milk allergy
- healthy control: healthy infants

SUMMARY:
Food allergy (FA) derives from a dysregulation of oral tolerance mechanisms. Studies suggest a crucial role for enteric microflora in oral tolerance development. An altered composition of intestinal microflora results in an unbalanced local and systemic immune response to food allergens. There are qualitative and quantitative differences in gut microbiota composition in children with food allergy. These findings support the concept that specific beneficial bacteria from human intestinal microflora, designated probiotics, could restore intestinal microflora homeostasis and prevent or treat FA.

ELIGIBILITY:
Inclusion Criteria:

* children with cow's milk allergy
* age 6-12 months

Exclusion Criteria:

* concomitant chronic systemic diseases
* congenital cardiac defects
* active tuberculosis
* autoimmune diseases
* immunodeficiency
* chronic inflammatory bowel diseases
* celiac disease, cystic fibrosis
* metabolic diseases
* malignancy
* chronic pulmonary diseases
* malformations of the gastrointestinal tract
* suspected eosinophilic esophagitis or eosinophilic enterocolitis
* suspected food-protein-induced enterocolitis syndrome.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Composition and function gut microbiota in children with cow milk allergy and healthy children | Change from baseline at 6 and 12 months

SECONDARY OUTCOMES:
Composition and function gut microbiota comparing cow milk allergy Italian and cow milk allergy children of other countries | Change from baseline at 6 and 12 months
Composition and function gut microbiota comparing healthy Italian and healthy children of other countries | Change from baseline at 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy